CLINICAL TRIAL: NCT06490757
Title: A Phase 2 Open-label Single-arm Trial of JAK1 Inhibitor for the Treatment of Large Inflammatory Hepatocellular Adenomas
Acronym: JAKIH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP220916
Record Dates: First submitted 2024-06-24; First posted 2024-07-08 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Hepatocellular Adenoma
Keywords: Hepatocellular adenoma; Inflammatory; JAK STAT pathway
MeSH Terms: conditions — Adenoma, Liver Cell | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ancillary study (Other): PET CT with 18 FDG will be performed in 12 patients in selected centers (Avicenne hospital, Beaujon hospital, Henri Mondor hospital, Bordeaux hospital, Paul brousse hospital, Saint Antoine hospital with nuclear medicine department available and should be done at baseline and 3 months (+/- one week).
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — An ancillary study will be performed in a subgroup of 12 patients to assess the variation of the results of PET-CT with 18FDG from baseline to 3 months. The variation of tumor features assessed by PET-CT with 18FDG after three months of treatment, will be assessed. The median value of the SUV max and tumor to non-tumor ratio of the SUV max value for each HCA lesion between the PET CT with 18FDG performed at baseline and after 3 months of treatment will be assessed.
  Other Names: fluorodésoxyglucose (18F)- Positron Emission Tomography (PET)

SUMMARY:
Hepatocellular adenomas (HCA) are tumors rare benign hepatic infections that develop on a liver normal and in young women taking a estrogen-based contraception. The main molecular subgroup of AHCs is the AHC subgroup inflammatory, which are associated with a risk of bleeding from the tumor and malignant transformation. Therefore, most of women with large inflammatory AHC (>5 cm) require liver resection which can be associated with morbidity and aesthetic problems, and rarely to mortality. On the basis of the knowledge of the molecular classification of AHCs humans and preclinical data testing the JAK1/2 inhibitors, we hypothesize that a short duration of treatment with the inhibitor of JAK1/2 (baricitinib) may be effective in patients with large inflammatory AHC size.

DETAILED DESCRIPTION:
Hepatocellular adenomas (HCA) are tumors rare benign hepatic infections that develop on a liver normal and in young women taking a estrogen-based contraception. The main molecular subgroup of AHCs is the AHC subgroup inflammatory, characterized by activation of the pathway JAK/STAT due to mutations in IL6ST, STAT3, FRK, JAK1 or GNAS, with inflammatory infiltrates at histology. Hepatocellular adenomas are associated with a risk of bleeding from the tumor and malignant transformation. Therefore, most of women with large inflammatory AHC (>5 cm) require liver resection which can be associated with morbidity and aesthetic problems, and rarely to mortality. On the basis of the knowledge of the molecular classification of AHCs humans and preclinical data testing the JAK1/2 inhibitors, we hypothesize that a short duration of treatment with the inhibitor of JAK1/2 (baricitinib) may be effective in patients with large inflammatory AHC size.

ELIGIBILITY:
Inclusion Criteria:

* Women (or male with inflammatory HCA considered as non resectable whatever the size of the HCA)
* Written informed consent for participation in study
* Histologically proven hepatocellular adenoma (confirmed by a centralized reviewing) with available FFPE
* At least one HCA of inflammatory subtype confirmed at histology and immunohistochemistry (CRP or SAA immunohistochemistry) by a centralized reviewing
* At least one HCA of more than 5 cm at imaging of inflammatory subtype (if the HCA of more than 5 cm is not the same HCA proved as inflammatory at histology this HCA should harbored the same imaging features than the HCA with available histology) for women.
* Diagnosed at histology over the last 5 years
* Absence of desire of pregnancy while treated by baricitinib and for at least 4 weeks following the last dose of investigational product
* Females of childbearing potential should have a contraception (without estrogen) when engaging in sexual intercourse with a male partner while treated by baricitinib and for at least 4 weeks following the last dose of investigational product. In case of oral contraception, patients should have been using it for a minimum of one month before the beginning of the treatment. A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Male when engaging in sexual intercourse with a female partner shoud have a contraception while treated by baricitinib and for at least 4 weeks following the last dose of investigational product A man is considered fertile after puberty unless permanently sterile by bilateral orchiectomy
* Past infection of Varicella zona Virus confirmed by serology or vaccine against Varicella zona Virus done more than 4 weeks before the inclusion
* Coverage for medical insurance

Exclusion criteria:

* < 18 years old and > 65 years old
* Pregnancy or breastfeeding woman
* Ongoing estrogen-based contraception at inclusion
* Patient on AME (state medical aid)
* Have a current or recent (<4 weeks prior to inclusion) clinically serious viral, bacterial, fungal, or parasitic infection (Note: For example, a recent viral upper respiratory tract infection or uncomplicated urinary tract infection should not be considered clinically serious).
* Have screening electrocardiogram (ECG) abnormalities that, in the opinion of the investigator or the sponsor, are clinically significant and indicate an unacceptable risk for the patient's participation in the study.
* Thrombocytopenia < 100 000/mm3
* Neutropenia < 1200/mm3
* Lymphopénia < 750/mm3
* Anemia < 9 g/dl
* Concomitant use of immunosuppressive treatment such as methotrexate, azathioprine, mycophenolate (at the exception of corticosteroid)
* Have received etanercept, infliximab, certolizumab, adalimumab, golimumab, or anakinra within 12 weeks of screening; tocilizumab, abatacept, ustekinumab, rituximab, belimumab, or any other B cell targeted therapies (approved or investigational) within 24 weeks of screening; or any other biologic therapy within 4 weeks of inclusion, whichever is longer.
* ASAT > 5 times upper fold of the normal or ALAT > 5 times upper fold of the normal or total bilirubin > upper 1.5 fold of the normal
* hepatic impairment defined by Child Pugh B or C
* Have evidence of active tuberculosis as documented by medical history, clinical symptoms, and abnormal chest x-ray at screening together with positive quantiferon or T spot test or positive culture
* Have evidence of latent TB (as documented by a positive quantiferon or T spot test, no clinical symptoms consistent with active TB, and a normal chest x-ray at screening, or as outlined below) unless patient completes at least 4 weeks of appropriate treatment prior to inclusion and agrees to complete the remainder of treatment while in the trial.
* Renal impairment with estimated creatinine clearance < 50 ml/mn (Cockroft and Gault formula)
* Have had any major surgery within 8 weeks prior to screening or will require major
* surgery during the study that, in the opinion of the investigator in consultation with the principal investigator, would pose an unacceptable risk to the patient.
* Past history of lymphoproliferative disease
* Past history of acute myocardial infection or unstable angina
* Past history of stroke (including transient ischemic attack)
* Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic BP (SBP), or > 100 mm Hg diastolic BP (DBP) despite optimal antihypertensive treatment
* Past history NYHA (New York Heart Association) class III or IV congestive heart failure
* Thromboembolic event within 6 months before inclusion
* current or past long-time smokers defined by more than 15 pack years
* Second or third atrioventricular block
* Active cancer
* Past history of cancer the 5 years before the inclusion with the following exception:
* -Patients with cervical carcinoma in situ that has been resected with no evidence of recurrence or metastatic disease for at least 3 years may participate in the study.
* -Patients with basal cell or squamous epithelial skin cancers that have been completely resected with no evidence of recurrence for at least 3 years may participate in the study.
* Have had symptomatic herpes zoster infection within 6 months prior to screening
* Have a past history of recurrent symptomatic zona (one single symptomatic zona that had occurred more than 6 months before the inclusion is not a contra-indication)
* Have a history of disseminated/complicated herpes zoster (for example, multidermatomal involvement, ophthalmic zoster, CNS involvement, or post-herpetic neuralgia).
* Have been exposed to a live vaccine within 12 weeks prior to planned inclusion or are expected to need/receive a live vaccine during the course of the study (with the exception of herpes zoster vaccination that must occur > 4 weeks prior to inclusion).
* Have active or chronic viral infection from hepatitis B virus (HBV, defined by positive aghbs), hepatitis C virus (HCV, defined by positive PCR), or human immunodeficiency virus (HIV, defined by positive serology).
* Patients under guardianship (tutelle/curatelle)
* Patient deprived of liberty under judicial or administrative decision.
* Participation in another interventional trial
* Hypersensitivity to the active substance (baricitinib) or to any of the excipients
* Past history of organ transplantation
* Surgery of the target IHCA required at diagnosis validated by a multidisciplinary tumor board during the screening process due to the following reason:
* Male with HCA accessible to liver resection (male not accessible to surgery based on a multidisciplinary tumor board evaluation could be included)
* Activation of the Wnt/B-catenin pathway at immunohistochemistry (diffuse positive glutamine synthase and/or nuclear translation of B-catenin) or mutations in exon 3 of CTNNB1 at molecular biology (except in this tumor is considered as unresectable) at the pathological reviewing
* Signs of malignant transformation in HCC (suspected by multidisciplinary tumor board based on imaging features or results of histology)
* Any other reasons validated by the multidisciplinary tumor board

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2028-09-02 (Estimated); Study Completion 2028-09-02 (Estimated)

PRIMARY OUTCOMES:
The principal outcome is to demonstrate that the combination of an experimental procedure to the standard of care lead to a significant decrease in size of large inflammatory HCA at imaging | 6 month
  The primary endpoint will be assessed at 6 months by comparing the liver MRI with contrast agent at baseline with the liver MRI with contrast agent at 6 months. An external independent reviewing will be performed separately by two radiologists that will classify the radiological response according to RECIST 1.1 criteria at 6 months in complete response, partial response, stable disease and progressive disease.

SECONDARY OUTCOMES:
Radiological response using RECIST 1.1 and at 3 months and 6 months | 3 months and 6 months
  Proportion of overall radiological response (partial and complete response), stable disease, and progressive disease using RECIST 1.1 criteria at 3 months and 6 months MRI
Decrease in size of the target lesions below 5 cm at 3 months and 6 months at imaging using RECIST 1.1 criteria | 3 months and 6 months
  Proportion of target lesions (inflammatory HCA > 5 cm) showing a decrease in size below 5 cm at 3 months and 6 months MRI using RECIST 1.1 thus modified RECIST criteria at MRI
Need for liver surgery of HCA at 6 months and 24 months (end of the follow-up) due to absence of sufficient decrease in size of the tumor under baricitinib | 6 months and 24 months
  Proportion patients treated by liver surgery for HCA at 6 months and the end of the 24 months follow-up
Incidence of adverse events related to the experimental treatment (baracitinib) | Inclusion at 24 month
  Adverse events within the 24 months of the study a) all adverse events b) occurrence of zona c) cancer d) major adverse cardiovascular events (MACE)
In patients with multiple HCA, radiological response using RECIST 1.1 at 3 months and 6 months focusing of HCA at the exclusion of the IHCA confirmed at histology | 3 months and 6 months
  In patients with multiple HCA, the proportion patients with complete response, partial response, stable disease and progressive disease focusing on other HCA excluding the inflammatory HCA confirmed at histology according to RECIST 1.1 criteria at MRI at 3 months and 6 months.
Symptomatic HCA bleeding during follow-up | follow-up (D15, M1, M3, M6, M12; M18 and M24)
  Proportion of symptomatic bleeding of HCA during follow-up
Incidence of malignant transformation of hepatocellular adenomas into hepatocellular carcinoma during the study | follow-up (D15, M1, M3, M6, M12; M18 and M24)
  Proportion of malignant transformation in HCC during follow-up at histology and confirmed by a multidisciplinary tumor board
Occurrence of increase in tumor size or number after discontinuation of baricitinib using RECIST 1.1 criteria during follow-up | baricitinib discontinuation (6 months) to 24 months
  Proportion of patients with a progressive disease between baricitinib discontinuation (6 months) and 24 months of follow-up using RECIST 1.1 criteria at imaging
Occurrence of increase in tumor size up to 5 cm after discontinuation of baricitinib using RECIST 1.1 criteria during follow-up | baricitinib discontinuation (6 months) to 24 months
  Proportion of patients with an increase in tumor size below 5 cm between baricitinib discontinuation (6 months) and 24 months at MRI
Incidence of post-operative adverse events in cases requiring hepatic surgery for hepatocellular adenoma during follow-up | follow-up (D15, M1, M3, M6, M12; M18 and M24)
  Proportion of post-operative adverse events (using the Dindo-Clavien Classification) if liver surgery is required during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles NAULT, PUPH, Principal Investigator — Assistance Publique des Hôpitaux de Paris (APHP)
Locations (1):
- NAULT, Bobigny, France

REFERENCES:
- [Background] Nault JC, Paradis V, Ronot M, Zucman-Rossi J. Benign liver tumours: understanding molecular physiology to adapt clinical management. Nat Rev Gastroenterol Hepatol. 2022 Nov;19(11):703-716. doi: 10.1038/s41575-022-00643-5. Epub 2022 Jul 14. PMID 35835851
- [Background] Zucman-Rossi J, Jeannot E, Nhieu JT, Scoazec JY, Guettier C, Rebouissou S, Bacq Y, Leteurtre E, Paradis V, Michalak S, Wendum D, Chiche L, Fabre M, Mellottee L, Laurent C, Partensky C, Castaing D, Zafrani ES, Laurent-Puig P, Balabaud C, Bioulac-Sage P. Genotype-phenotype correlation in hepatocellular adenoma: new classification and relationship with HCC. Hepatology. 2006 Mar;43(3):515-24. doi: 10.1002/hep.21068. PMID 16496320
- [Background] European Association for the Study of the Liver (EASL). EASL Clinical Practice Guidelines on the management of benign liver tumours. J Hepatol. 2016 Aug;65(2):386-98. doi: 10.1016/j.jhep.2016.04.001. Epub 2016 Apr 13. No abstract available. PMID 27085809
- [Background] Dokmak S, Paradis V, Vilgrain V, Sauvanet A, Farges O, Valla D, Bedossa P, Belghiti J. A single-center surgical experience of 122 patients with single and multiple hepatocellular adenomas. Gastroenterology. 2009 Nov;137(5):1698-705. doi: 10.1053/j.gastro.2009.07.061. Epub 2009 Aug 5. PMID 19664629
- [Background] Rebouissou S, Amessou M, Couchy G, Poussin K, Imbeaud S, Pilati C, Izard T, Balabaud C, Bioulac-Sage P, Zucman-Rossi J. Frequent in-frame somatic deletions activate gp130 in inflammatory hepatocellular tumours. Nature. 2009 Jan 8;457(7226):200-4. doi: 10.1038/nature07475. Epub 2008 Nov 19. PMID 19020503
- [Background] Bayard Q, Caruso S, Couchy G, Rebouissou S, Bioulac Sage P, Balabaud C, Paradis V, Sturm N, de Muret A, Guettier C, Bonsang B, Copie C, Letouze E, Calderaro J, Imbeaud S, Nault JC, Zucman-Rossi J. Recurrent chromosomal rearrangements of ROS1, FRK and IL6 activating JAK/STAT pathway in inflammatory hepatocellular adenomas. Gut. 2020 Sep;69(9):1667-1676. doi: 10.1136/gutjnl-2019-319790. Epub 2020 Jan 6. PMID 31907296
- [Background] Poussin K, Pilati C, Couchy G, Calderaro J, Bioulac-Sage P, Bacq Y, Paradis V, Leteurtre E, Sturm N, Ramos J, Guettier C, Bardier-Dupas A, Boulai A, Wendum D, Selves J, Izard T, Nault JC, Zucman-Rossi J. Biochemical and functional analyses of gp130 mutants unveil JAK1 as a novel therapeutic target in human inflammatory hepatocellular adenoma. Oncoimmunology. 2013 Dec 1;2(12):e27090. doi: 10.4161/onci.27090. Epub 2014 Jan 3. PMID 24501689
- [Background] Simpson EL, Lacour JP, Spelman L, Galimberti R, Eichenfield LF, Bissonnette R, King BA, Thyssen JP, Silverberg JI, Bieber T, Kabashima K, Tsunemi Y, Costanzo A, Guttman-Yassky E, Beck LA, Janes JM, DeLozier AM, Gamalo M, Brinker DR, Cardillo T, Nunes FP, Paller AS, Wollenberg A, Reich K. Baricitinib in patients with moderate-to-severe atopic dermatitis and inadequate response to topical corticosteroids: results from two randomized monotherapy phase III trials. Br J Dermatol. 2020 Aug;183(2):242-255. doi: 10.1111/bjd.18898. Epub 2020 Mar 5. PMID 31995838
- [Background] Nault JC, Couchy G, Balabaud C, Morcrette G, Caruso S, Blanc JF, Bacq Y, Calderaro J, Paradis V, Ramos J, Scoazec JY, Gnemmi V, Sturm N, Guettier C, Fabre M, Savier E, Chiche L, Labrune P, Selves J, Wendum D, Pilati C, Laurent A, De Muret A, Le Bail B, Rebouissou S, Imbeaud S; GENTHEP Investigators; Bioulac-Sage P, Letouze E, Zucman-Rossi J. Molecular Classification of Hepatocellular Adenoma Associates With Risk Factors, Bleeding, and Malignant Transformation. Gastroenterology. 2017 Mar;152(4):880-894.e6. doi: 10.1053/j.gastro.2016.11.042. Epub 2016 Dec 7. PMID 27939373
- [Background] Bioulac-Sage P, Rebouissou S, Thomas C, Blanc JF, Saric J, Sa Cunha A, Rullier A, Cubel G, Couchy G, Imbeaud S, Balabaud C, Zucman-Rossi J. Hepatocellular adenoma subtype classification using molecular markers and immunohistochemistry. Hepatology. 2007 Sep;46(3):740-8. doi: 10.1002/hep.21743. PMID 17663417
- [Background] Demory A, Peron JM, Calderaro J, Selves J, Mokrane FZ, Amaddeo G, Paradis V, Ziol M, Sutter O, Blaise L, Ganne-Carrie N, Vilgrain V, Cauchy F, Zucman-Rossi J, Ronot M, Nault JC. Body weight changes and duration of estrogen exposure modulate the evolution of hepatocellular adenomas after contraception discontinuation. Hepatology. 2023 Feb 1;77(2):430-442. doi: 10.1002/hep.32734. Epub 2022 Sep 11. PMID 35980227
- [Background] Bioulac-Sage P, Laumonier H, Couchy G, Le Bail B, Sa Cunha A, Rullier A, Laurent C, Blanc JF, Cubel G, Trillaud H, Zucman-Rossi J, Balabaud C, Saric J. Hepatocellular adenoma management and phenotypic classification: the Bordeaux experience. Hepatology. 2009 Aug;50(2):481-9. doi: 10.1002/hep.22995. PMID 19585623
- [Background] Vernuccio F, Ronot M, Dioguardi Burgio M, Cauchy F, Choudhury KR, Dokmak S, Soubrane O, Valla D, Zucman-Rossi J, Paradis V, Vilgrain V. Long-term Evolution of Hepatocellular Adenomas at MRI Follow-up. Radiology. 2020 May;295(2):361-372. doi: 10.1148/radiol.2020191790. Epub 2020 Mar 17. PMID 32181728
- [Background] van Rosmalen BV, Furumaya A, Klompenhouwer AJ, Tushuizen ME, Braat AE, Reinten RJ, Ligthart MAP, Haring MPD, de Meijer VE, van Voorthuizen T, Takkenberg RB, Dejong CHC, de Man RA, IJzermans JNM, Doukas M, van Gulik TM, Verheij J; Dutch Benign Liver Tumor Group and the PALGA group. Hepatocellular adenoma in men: A nationwide assessment of pathology and correlation with clinical course. Liver Int. 2021 Oct;41(10):2474-2484. doi: 10.1111/liv.14989. Epub 2021 Jul 8. PMID 34155783
- [Background] Von Hoff DD, LoRusso PM, Rudin CM, Reddy JC, Yauch RL, Tibes R, Weiss GJ, Borad MJ, Hann CL, Brahmer JR, Mackey HM, Lum BL, Darbonne WC, Marsters JC Jr, de Sauvage FJ, Low JA. Inhibition of the hedgehog pathway in advanced basal-cell carcinoma. N Engl J Med. 2009 Sep 17;361(12):1164-72. doi: 10.1056/NEJMoa0905360. Epub 2009 Sep 2. PMID 19726763
- [Background] Gross AM, Wolters PL, Dombi E, Baldwin A, Whitcomb P, Fisher MJ, Weiss B, Kim A, Bornhorst M, Shah AC, Martin S, Roderick MC, Pichard DC, Carbonell A, Paul SM, Therrien J, Kapustina O, Heisey K, Clapp DW, Zhang C, Peer CJ, Figg WD, Smith M, Glod J, Blakeley JO, Steinberg SM, Venzon DJ, Doyle LA, Widemann BC. Selumetinib in Children with Inoperable Plexiform Neurofibromas. N Engl J Med. 2020 Apr 9;382(15):1430-1442. doi: 10.1056/NEJMoa1912735. Epub 2020 Mar 18. PMID 32187457
- [Background] McLornan DP, Pope JE, Gotlib J, Harrison CN. Current and future status of JAK inhibitors. Lancet. 2021 Aug 28;398(10302):803-816. doi: 10.1016/S0140-6736(21)00438-4. PMID 34454676
- [Background] Taylor PC, Keystone EC, van der Heijde D, Weinblatt ME, Del Carmen Morales L, Reyes Gonzaga J, Yakushin S, Ishii T, Emoto K, Beattie S, Arora V, Gaich C, Rooney T, Schlichting D, Macias WL, de Bono S, Tanaka Y. Baricitinib versus Placebo or Adalimumab in Rheumatoid Arthritis. N Engl J Med. 2017 Feb 16;376(7):652-662. doi: 10.1056/NEJMoa1608345. PMID 28199814
- [Background] Petri M, Bruce IN, Dorner T, Tanaka Y, Morand EF, Kalunian KC, Cardiel MH, Silk ME, Dickson CL, Meszaros G, Zhang L, Jia B, Zhao Y, McVeigh CJ, Mosca M. Baricitinib for systemic lupus erythematosus: a double-blind, randomised, placebo-controlled, phase 3 trial (SLE-BRAVE-II). Lancet. 2023 Mar 25;401(10381):1011-1019. doi: 10.1016/S0140-6736(22)02546-6. Epub 2023 Feb 24. PMID 36848919
- [Background] Marconi VC, Ramanan AV, de Bono S, Kartman CE, Krishnan V, Liao R, Piruzeli MLB, Goldman JD, Alatorre-Alexander J, de Cassia Pellegrini R, Estrada V, Som M, Cardoso A, Chakladar S, Crowe B, Reis P, Zhang X, Adams DH, Ely EW; COV-BARRIER Study Group. Efficacy and safety of baricitinib for the treatment of hospitalised adults with COVID-19 (COV-BARRIER): a randomised, double-blind, parallel-group, placebo-controlled phase 3 trial. Lancet Respir Med. 2021 Dec;9(12):1407-1418. doi: 10.1016/S2213-2600(21)00331-3. Epub 2021 Sep 1. PMID 34480861
- [Background] Sanchez GAM, Reinhardt A, Ramsey S, Wittkowski H, Hashkes PJ, Berkun Y, Schalm S, Murias S, Dare JA, Brown D, Stone DL, Gao L, Klausmeier T, Foell D, de Jesus AA, Chapelle DC, Kim H, Dill S, Colbert RA, Failla L, Kost B, O'Brien M, Reynolds JC, Folio LR, Calvo KR, Paul SM, Weir N, Brofferio A, Soldatos A, Biancotto A, Cowen EW, Digiovanna JJ, Gadina M, Lipton AJ, Hadigan C, Holland SM, Fontana J, Alawad AS, Brown RJ, Rother KI, Heller T, Brooks KM, Kumar P, Brooks SR, Waldman M, Singh HK, Nickeleit V, Silk M, Prakash A, Janes JM, Ozen S, Wakim PG, Brogan PA, Macias WL, Goldbach-Mansky R. JAK1/2 inhibition with baricitinib in the treatment of autoinflammatory interferonopathies. J Clin Invest. 2018 Jul 2;128(7):3041-3052. doi: 10.1172/JCI98814. Epub 2018 Jun 11. PMID 29649002
- [Background] Morand EF, Vital EM, Petri M, van Vollenhoven R, Wallace DJ, Mosca M, Furie RA, Silk ME, Dickson CL, Meszaros G, Jia B, Crowe B, de la Torre I, Dorner T. Baricitinib for systemic lupus erythematosus: a double-blind, randomised, placebo-controlled, phase 3 trial (SLE-BRAVE-I). Lancet. 2023 Mar 25;401(10381):1001-1010. doi: 10.1016/S0140-6736(22)02607-1. Epub 2023 Feb 24. PMID 36848918
- [Background] King B, Ohyama M, Kwon O, Zlotogorski A, Ko J, Mesinkovska NA, Hordinsky M, Dutronc Y, Wu WS, McCollam J, Chiasserini C, Yu G, Stanley S, Holzwarth K, DeLozier AM, Sinclair R; BRAVE-AA Investigators. Two Phase 3 Trials of Baricitinib for Alopecia Areata. N Engl J Med. 2022 May 5;386(18):1687-1699. doi: 10.1056/NEJMoa2110343. Epub 2022 Mar 26. PMID 35334197
- [Background] Ytterberg SR, Bhatt DL, Mikuls TR, Koch GG, Fleischmann R, Rivas JL, Germino R, Menon S, Sun Y, Wang C, Shapiro AB, Kanik KS, Connell CA; ORAL Surveillance Investigators. Cardiovascular and Cancer Risk with Tofacitinib in Rheumatoid Arthritis. N Engl J Med. 2022 Jan 27;386(4):316-326. doi: 10.1056/NEJMoa2109927. PMID 35081280
- [Background] Gregory J, Dioguardi Burgio M, Corrias G, Vilgrain V, Ronot M. Evaluation of liver tumour response by imaging. JHEP Rep. 2020 Apr 28;2(3):100100. doi: 10.1016/j.jhepr.2020.100100. eCollection 2020 Jun. PMID 32514496